CLINICAL TRIAL: NCT03625206
Title: Cognitive Bias Modification Training in Adolescents Who Have Experienced Adversity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Psychiatry, London (Other)
Collaborators: Banaras Hindu University (Other); Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Jennifer Lau, Principal Investigator, Institute of Psychiatry, London
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PAHBABR
Record Dates: First submitted 2018-07-04; First posted 2018-08-10 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Child Abuse; Child Neglect; Victimization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are told that they will be allocated to one of two intervention conditions, one which may be more effective than the other in challenging negative thought patterns. Outcome assessors are blind to the status of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive bias modification training (Experimental): Participants will receive 5 training sessions, each session including attention bias modification and interpretation bias modification training modules
  Interventions: Behavioral: Cognitive bias modification training
- Control training (Placebo Comparator): Participants will receive 5 sessions that involve exercises that are matched to the task demands of the attention bias modification and interpretation bias modification training modules
  Interventions: Behavioral: Control training

INTERVENTIONS:
Behavioral: Cognitive bias modification training — These training sessions aim to modify a selective attention bias towards threat and a tendency to interpret ambiguous situations in threatening ways
  Arms: Cognitive bias modification training
Behavioral: Control training — These exercises are matched to the task demands of the modules of cognitive bias modification training
  Arms: Control training

SUMMARY:
Adolescents who have experienced adversity (childhood maltreatment and other forms of broader victimisation experiences) will be randomly allocated to receive a 5-session cognitive bias modification training (with attention and interpretation bias modification modules) or a control condition. Outcome measures include measures of cognitive biases and symptoms of psychopathology; in addition, in a subset of adolescents, brain activity data will be acquired. All adolescents will complete a feedback form, upon which acceptability of the intervention will be assessed.

DETAILED DESCRIPTION:
Up to 80 adolescents aged 12-18 years who have experienced adversity (childhood maltreatment and other forms of broader victimisation experiences) from India and Nepal will be randomly allocated to receive a 5-session cognitive bias modification training (with attention and interpretation bias modification modules) or a control condition over a 2-week period.

Pre and post-assessment measures include measures of attention and interpretation biases and symptoms of internalising and externalising psychopathology. In addition, in a subset of adolescents, brain activity data acquired using EEG will be acquired either during resting or viewing emotional face stimuli. Data from these measures will be used to generate effect sizes of changes for each group as well as being used in a limited number of significance-testing analysis. All adolescents will complete a feedback form, upon which acceptability of the intervention will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-18 years
* Adolescents who have experienced adversity (abuse, neglect) or broader victimisation experiences (conventional crime)

Exclusion Criteria:

* Adolescents who have difficulty reading or understanding what is being read to them
* Adolescents who are currently at-risk for self-harm
* Adolescents who are currently experiencing psychotic symptoms
* Adolescents who are currently experiencing high-level trauma symptoms

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2020-05-17 (Actual); Study Completion 2020-05-17 (Actual)

PRIMARY OUTCOMES:
Attention biases for threatening stimuli | Immediately after the intervention (post-intervention)
  The investigators will use an experimental measure (a visual search task) that uses reaction times (RTs) to different experimental conditions to index the degree to which attention is captured by a threatening over a non-threatening stimulus.
Interpretation biases for threatening explanations | Immediately after the intervention (post-intervention)
  The investigators will use an experimental measure (an ambiguous scenarios task) that uses ratings to different experimental trials to index the degree to which individuals endorse threatening over benign interpretations

SECONDARY OUTCOMES:
Symptoms of emotional, behavioural and social problems | Immediately after the intervention (post-intervention)
  5 subscales of the Strength and Difficulties questionnaire
Acceptability of intervention | Immediately after the intervention (post-intervention)
  The investigators have developed a 19-item self-report feedback, comprising quantitative ratings and qualitative responses. Across eleven items, young people rate on a 4-point Likert scale whether they found the training useful, satisfying, engaging, realistic, whether it impacted anxiety, mood, coping strategies, and other difficulties , and whether they would feel motivated to complete the sessions, including without a researcher present. Higher scores reflect greater endorsement. Each of these items will be reported separately rather than used to create composite scores. There are also 8 open ended questions for young people to leave their feedback on aspects they found helpful, unhelpful, liked, disliked, improvements they would want, and other general comments.
Event related potentials to emotional face presentations during Electroencephalogram (EEG) experiment | Immediately after the intervention (post-intervention)
  P1, N1, P2, N2, P3 event-related potentials during face presentation

CONTACTS AND LOCATIONS:
Locations (2):
- Psychology Department, Varanasi, India
- Psychology Department, Tribuwan University, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
All data will be anonymised such that each participant will be associated with a unique identification (ID) number. These will be uploaded to data repository sites once data collection, analysis and dissemination is completed
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Only once data collection, analysis and dissemination is completed

REFERENCES:
- [Derived] Dhakal S, Gupta S, Sharma NP, Upadhyay A, Oliver A, Sumich A, Kumari V, Niraula S, Pandey R, Lau JYF. Can we challenge attention and interpretation threat biases in rescued child labourers with a history of physical abuse using a computerised cognitive training task? Data on feasibility, acceptability and target engagement. Behav Res Ther. 2023 Mar;162:104267. doi: 10.1016/j.brat.2023.104267. Epub 2023 Jan 29. PMID 36780810